CLINICAL TRIAL: NCT02990832
Title: Diabetes Foot Care Clinical Pathway Project - Exciton Technologies Inc
Acronym: DFCCP-Exciton
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was deemed unfeasible to complete.
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Exciton Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Catherine Chan, Professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AICE-201500872
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exciton (Experimental): Treatment of diabetic foot ulcer with Exciton Exsalt wound dressing
  Interventions: Device: Exciton

INTERVENTIONS:
Device: Exciton — Exsalt® Wound Dressings will be applied by the physician/nursing staff.
  The test product, exsalt® Wound Dressings (0.4 mg Ag/cm2) will be applied after wound cleansing or debridement if required.
  Dressings will be changed weekly, either at the out-patient facility or at home with provided dressings. At regular intervals throughout the study, as per the existing Diabetes Foot Care Clinical Care Pathway, wound assessment including size determination, Exsalt Wound Assessment Form, any adverse events will be reported, with tracing and/or photography included where available.
  Maximum treatment course will be 28 days (end of study) or until wound closure.

SUMMARY:
In 2011, the premiers of all Canadian provinces and territories selected diabetes foot care as 1 of 3 significant targets for pan-provincial action. Of 210,000 people with diabetes in Alberta, 5,250 will seek treatment of a foot ulcer annually. In Alberta in 2014-15 there were 425 lower limb amputations (LLA). Moreover, there is a tremendous reduction in quality of life of the patients and attendant negative effects on their families. The 5-year mortality rate after new-onset diabetic foot ulcer is 43-55% and as high as 74% for patients undergoing LLA (CIHI, 2013). The Diabetes Foot Care Clinical Pathway Project (DFCCPP) aims to optimize methods of early detection and treatment of foot ulcers in an effort to reduce LLA by 50% by implementing High Risk Foot Teams (HRFTs) across the province starting with 3 Pilot sites. Existing staff with expertise and knowledge in diabetic foot care will assess and treat patients with moderate and high-risk findings.

In conjunction with the DFCCPP, the efficacy of a technological advancement developed by an Alberta-based small-to-medium enterprise (SME) to improve diabetic foot outcomes will be evaluated. Exsalt® SD7 Wound Dressings (Exciton Technologies, Edmonton, AB) have been demonstrated in-vitro and in-vivo to provide rapid and effective antibacterial activity in an easy-to-use format, thus creating an enhanced wound healing environment while supporting patient quality of life.

The objective of the proposed work is twofold, namely 1) to quantify clinical efficacy of exsalt® Wound Dressings on locally infected diabetic foot ulcers not progressing to healing under the current standard of care: evaluating key indicators of infection, Infectious Diseases Society of America (IDSA) wound classification, and wound size; identifying benefits to foot ulcer healing and 2) to evaluate subjective patient outcomes: satisfaction, perceived benefit, compliance. Evaluating the benefits of utilization of the Exciton exsalt® Wound Dressings when combined with the DFCCP.

DETAILED DESCRIPTION:
2 Background Information

2.1 Device Description

Exsalt® Wound Dressings (Test Dressings) contain oxidized silver oxysalts deposited throughout a non-woven polyester/High density polyethylene non-adherent dressing. Silver in the exsalt® Wound Dressings inhibits microbial growth in the dressing. The concentration of the silver and oxidized silver species on the dressing is 0.4 mg/cm2 (2.5% w/w). The exsalt® dressings have been shown to be effective in vitro against Staphylococcus aureus, Escherichia coli, Pseudomonas aeruginosa, and Enterococcus faecalis. Exsalt® Wound Dressings maintain their antibacterial activity for up to 7 days against Pseudomonas aeruginosa and Staphylococcus aureus.

Exsalt® Wound Dressings are indicated for the management of partial and full thickness wounds, including decubitus ulcers, venous stasis ulcers, diabetic ulcers, first and second degree burns, grafts and donor sites, or other acute or chronic wounds. The dressing may be used over debrided and grafted wounds.

2.2 Study History

The Canadian Institute of Health Information estimates that foot wounds (with diabetes as the leading cause) are present in 4% of all hospital inpatients, 7% of homecare clients and 10% of long-term care residents (CIHI, 2013). Ulcerations are a critical event in the loss of limbs or amputation as they create an avenue for infection and may exacerbate necrotic tissue and ischemia. Of 210,000 people with diabetes in Alberta, 5,250 will seek treatment of a foot ulcer annually. In Alberta in 2014-15 there were 425 LLA performed on 309 diabetic patients representing an increase of 89 LLA over 2010-11.

The 5-year mortality rate after new-onset diabetic foot ulcer is 43-55% and as high as 74% for patients undergoing LLA (Ollendorf et al, 1998). Moreover, there is a tremendous reduction in quality of life of the patients and negative effects on their families. The Diabetes Foot Care Clinical Pathway Project (DFCCPP) aims to optimize methods of early detection and treatment of foot ulcers in an effort to reduce LLA by 50% and improve patient's quality of life. Therefore, there is a need for an effective tool for the prevention and management of local infection in diabetic foot ulcers.

2.3 Device History

Exsalt® wound dressings have to date been formally evaluated (including clinical studies and post-market surveillance) on over 125 patients throughout North America and Europe. In these studies, many wound etiologies were investigated including: venous leg ulcers, diabetic ulcers, diabetic neuropathic ulcers, post-surgical wounds, wounds resulting from trauma, skin tears, pressure ulcers, burn wounds, and chronic non-healing ulcers. The formal clinical evaluations investigated the safety and efficacy of the Exsalt® wound dressing as a device. Data and feedback generated supported wound healing, with increased granulation tissue and lessened pain, odor, and signs of infection (Thomason et al, 2016; Lemire et al, 2015). The wound dressing was shown to support progression to wound closure or wound healing without signs of toxicity or side-effects.

2.4 Risk Summary

Precautions need to be taken when using exsalt® Wound Dressing as it should not be used on patients with a known sensitivity to silver; is not compatible with oil-based products, such as petrolatum; is not compatible with magnetic resonance imaging (MRI) procedures; should be removed prior to administering radiation therapy; and should not come in contact with electrodes and conductive gels during electronic measurements (e.g. EEG, ECG).

Additionally, frequent or prolonged use of Exsalt® wound dressings may result in permanent discoloration of skin.

2.5 Benefit Summary

Benefits of this product vs. other silver antimicrobials include rapid and sustained bactericidal activity; broad spectrum of activity; minimized pain; reduced staining of skin; non-toxicity to human tissue; decreased likelihood of resistance; cost-effectiveness as it requires less silver.

2.6 Good Clinical Practice and Regulatory Requirements

2.6.1 Regulatory Requirements: Exsalt® Wound Dressing

Exsalt® Wound Dressings exsalt® SD7 and exsalt® T7 have been licensed in Canada by Health Canada as of January 2011 and March 2012, respectively. Exsalt® wound dressing is "indicated for the management of partial and full thickens wounds such as decubitus ulcers, venous stasis ulcers, diabetic ulcers, 1st and 2nd degree burns, grafts and donor sites' or other acute or chronic wounds."

3 Study Objectives & Purpose

The purpose of this pilot study is to evaluate the effectiveness of the Exciton exsalt® Wound Dressings when combined with the DFCCP in patients with locally infected diabetic foot ulcers. The objective of the proposed work is twofold, namely 1) to quantify the effectiveness of exsalt® Wound Dressings on locally infected diabetic foot ulcers not progressing to healing under the current standard of care: evaluating IDSA wound classification, pain, wound size, and signs and symptoms of infection through a one-arm prospective repeated measures pilot study and 2) to compile subjective patient outcomes: satisfaction, perceived benefit, compliance. Evaluating the benefits of utilization of the Exciton exsalt® Wound Dressings when combined with the DFCCP.

Specifically, the following work and objectives are proposed:

1. A prospective, single-arm, repeated measures study to pilot the use of Exsalt® wound dressing in chronic wounds within an outpatient clinical setting; evaluate the benefits of utilization of exsalt® Wound Dressings within the DFCCPP.
2. Repeated measures evaluating and reporting wound infection classification (IDSA), pain score, wound size, and key indicators of infection; pre and post-intervention. Quantifying the impact of the intervention to diabetic foot ulcer local infection, healing, and associated pain. Qualifying subjective patient outcomes including satisfaction, benefit, and compliance. Incidence of safety and adverse events will be reported within the scope of this pilot study.

3.1 Research Questions

The research proposed here is designed to address the following questions:

1. What is the impact (monitoring key indicators of infection, wound size, and wound classification) of the application of the exsalt® Wound Dressing utilized as a primary dressing for up to four weeks in outpatients with diabetic foot ulcers that have a mild local infection and are non-responsive using standard-of-care.?
2. What is the clinical utility of the use of the Exsalt® wound dressing from the perspective of clinical staff and patients?
3. What are the benefits of utilization of the Exciton exsalt® Wound Dressings when combined with the DFCCP?

4 Pilot Study Design

4.1 Study type

A prospective, single-arm, repeated measures study pilot study will be coordinated by the DON-SCN on the use of exsalt® Wound Dressings in mildly infected chronic diabetic foot ulcer wounds within three outpatient clinical settings; evaluating pre and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus according to definitions outlined by the American Diabetes Association
* Presenting with a localized mild infection of the ulcer as listed in the IDSA Clinical Practice Guideline for the Diagnosis and Treatment of Diabetic Foot Infections (Table 1); exceeding 0.5 cm2 in area after appropriate debridement
* Diagnosis of mild infection must be confirmed immediately following debridement at Baseline
* Subject must agree to adhere to all protocol procedures and must be willing and able to provide written informed consent.
* Correction or optimization of underlying medical problems (e.g. diabetes or systemic infection).
* Wound has been identified as stalled or persistent non-healing under current standard-of-care; showing no progression in 2 weeks as per IDSA guidelines

Exclusion Criteria:

* Use of systemic antibiotics within the previous 2 weeks
* Known silver sensitivity
* Current use of enzymatic debridement
* Wounds where best practice wound bed preparation is not available or applicable (eg, wound with diminutive oxygen supply would be contraindicated for debridement.
* No palpable dorsalis pedis or posterior tibial pulse or a pedal systolic pressure (Doppler) of ≤ 40 mm Hg
* Evidence of systemic infection (fever, chills, hypotension)/sepsis
* Non-study systemic or anti-infective topical agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Infection assessed as per Infectious Disease Society of America (IDSA) guidelines | 28 days
  Assessed as per Infectious Disease Society of America (IDSA) guidelines

SECONDARY OUTCOMES:
Pain assessed with Ordinal scale | 28 days
  Ordinal scale, 0=none, 3=severe
Wound volume | 28 days
  Wound area multiplied by wound depth (cubic centimetres)
Safety and complications (incidence of adverse events) | 28 days
  The principal measure of safety will be the incidence of adverse events reported during the study. Adverse events from patients will be noted and thoroughly documented. Patients who experience adverse events may or may not be withdrawn from the study, depending on the nature and timing of the event; study investigators will review and assess each adverse event on a case-by-case basis. Data for safety assessments will be collected from all completed adverse events reports.

IPD SHARING:
Plan to Share IPD: No